CLINICAL TRIAL: NCT00142519
Title: Translational Studies in Analgesic Pharmacology: Analgesic Synergy in Clinical Pain. A Phase 2 Study Comparing a Single Dose of a 1:1 Combination of Methadone and Morphine With Morphine Alone in Patients With Post-operative Pain.
Brief Title: Comparison of A Single Dose Combination of Methadone and Morphine With Morphine Alone for Treating Post-operative Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05-025
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Results first posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2018-08

CONDITIONS: Pain
Keywords: Pain; Analgesics; Retroperitoneal lymph node dissection
MeSH Terms: conditions — Pain | interventions — Methadone; Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator): methadone
  Interventions: Drug: Methadone
- 2 (Experimental): methadone and morphine
  Interventions: Drug: methadone and morphine

INTERVENTIONS:
Drug: Methadone — Upon the 1st request for analgesic medication morphine 2 mg, upon the 2nd request for analgesic medication morphine 2 mg
  Arms: 1
Drug: methadone and morphine — Upon the 1st request for analgesic medication morphine 2 mg, upon the 2nd request for analgesic medication morphine 1 mg and methadone 1 mg
  Arms: 2

SUMMARY:
This is a randomized Phase II study testing the effectiveness of the combination of morphine and methadone versus morphine alone in relieving pain. A second goal is to further evaluate any side effects of the combination of morphine and methadone.

DETAILED DESCRIPTION:
Rationale: Experimental data demonstrates a profound analgesic synergy between morphine and methadone when co-administered systemically in mice. If this type of synergy can be demonstrated in clinical pain, it will be a relatively unique example of translating concepts of fundamental aspects of opioid actions seen in the laboratory to the clinical area, and provide a basis for offering new and scientifically- based analgesic regimens. This may provide better pain relief with less opioid related side effects in clinical practice.

Purpose:

This is a randomized, double blind, parallel arm Phase II study comparing a single dose of 1:1 combination of methadone and morphine with morphine alone in patients with post-operative pain.

* The primary objective of this randomized, double blind, parallel arm Phase II study is to compare the analgesic effects of a combination of morphine and methadone with morphine alone to determine synergistic activity of mu opioid analgesics in patients with post-operative pain.
* A second goal is to further evaluate any side effects of the combination of morphine and methadone.

ELIGIBILITY:
Inclusion Criteria:

* Retroperitoneal lymph node dissection
* Planned post-operative analgesia with PCA at 1 mg continuous infusion and 1 mg every 10 minutes
* 18 years of age or older
* English-speaking
* Give informed consent to participate in this study

Exclusion Criteria:

* Known hypersensitivity to methadone or morphine
* Patients with past or present history of substance abuse
* Patients with a history of methadone treatment
* Patients with a history of chronic pain requiring daily analgesic use for more than 3 months
* Patients treated with opioids within one month from the scheduled surgery
* Creatinine clearance less than 50 mg/kg (using Cockcroft-Gault Equation).
* Neurologic or psychiatric disease sufficient, in the doctor's opinion, to compromise data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-03 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Moryl, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Methadone: methadone
  Methadone: Upon the 1st request for analgesic medication morphine 2 mg, upon the 2nd request for analgesic medication morphine 2 mg
- Methadone and Morphine: methadone and morphine
  methadone and morphine: Upon the 1st request for analgesic medication morphine 2 mg, upon the 2nd request for analgesic medication morphine 1 mg and methadone 1 mg
Period: Overall Study
Arm/Group | Methadone | Methadone and Morphine
Started | 25 | 25
Completed | 7 | 9
Not Completed | 18 | 16
Not completed — Not Treated | 7 | 9
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 10 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methadone | Methadone and Morphine | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Full Range); unit: years] | 34.9 [19 to 67] | 31.6 [18 to 55] | 33.2 [18 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 25 | 25 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 23 | 23 | 46
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: The Primary Goal of This Study is to Compare the Analgesic Effects of a Combination of Morphine and Methadone With Morphine Alone to Determine Synergistic Activity of mu Opioid Analgesics in Patients With Post-operative Pain.
Time Frame: Time to the third request for the pain medication
Population: Data not collected
Arm/Group | Methadone | Methadone and Morphine
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: To Determine if There Are Any Side Effects From the Combination of Morphine and Methadone When Given Together.
Time Frame: assessed every 10 minutes
Population: Data not collected
Arm/Group | Methadone | Methadone and Morphine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Methadone | Methadone and Morphine
All-Cause Mortality (participants affected / at risk) | 2/25 | 2/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2008-10-14): https://cdn.clinicaltrials.gov/large-docs/19/NCT00142519/Prot_SAP_000.pdf